CLINICAL TRIAL: NCT00007982
Title: CAMP 004A - Phase 2 Study Of Intensive Chemotherapy (BET) For Selected Categories Of Malignant Central Nervous System Tumor
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplant in Treating Patients With Central Nervous System Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068360; CPMC-IRB-8445; CPMC-CAMP-004A; NCI-G00-1881
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2007-07

CONDITIONS: Brain and Central Nervous System Tumors; Head and Neck Cancer; Lymphoma
Keywords: recurrent adult brain tumor; adult medulloblastoma; adult oligodendroglioma; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; adult anaplastic astrocytoma; adult central nervous system germ cell tumor; primary central nervous system non-Hodgkin lymphoma; adult anaplastic oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms; Lymphoma; Brain Neoplasms; Medulloblastoma; Oligodendroglioma; Esthesioneuroblastoma, Olfactory; Astrocytoma | interventions — Filgrastim; Carmustine; Cisplatin; Cyclophosphamide; Etoposide; Thiotepa; Chemotherapy, Adjuvant; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: thiotepa
Procedure: adjuvant therapy
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well chemotherapy and peripheral stem cell transplant work in treating patients with central nervous system cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with central nervous system malignancies treated with intensive chemotherapy supported by autologous peripheral blood stem cell transplantation following surgical resection and/or radiotherapy.
* Determine the disease-free survival and overall survival of this patient population treated with these regimens.
* Determine the toxicity of this high-dose chemotherapy regimen in these patients.
* Assess the quality of life of these patients following these treatment regimens.

OUTLINE: Patients with anaplastic astrocytoma, esthesioneuroblastoma, germ cell tumor, or primary neuroectodermal tumor undergo initial surgical resection followed by conventional or stereotactic radiotherapy. Patients with germ cell or primary neuroectodermal tumors also receive 4 courses of standard chemotherapy comprising cyclophosphamide, etoposide, and cisplatin prior to high-dose chemotherapy.

All patients undergo peripheral blood stem cell or bone marrow harvest followed by high-dose chemotherapy consolidation. Patients receive thiotepa IV 3 times daily on days -7 to -3, carmustine IV over 1 hour on days -6 to -3, and etoposide IV over 5 hours on days -6 to -3. Patients then undergo transplantation on day 0. Filgrastim (G-CSF) is administered concurrently with stem cell harvesting and transplantation.

Patients with recurrent oligodendroglioma or CNS lymphoma who have not received radiotherapy at diagnosis undergo conventional radiotherapy 6 weeks after completion of high-dose chemotherapy.

Patients are followed every 2-3 months for 1 year and then annually for 5 years. Quality of life is assessed at follow-up.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant tumors

  * Anaplastic astrocytoma
  * Oligodendroglioma
  * Germ cell tumor
  * Medulloblastoma
  * Primary neuroectodermal tumor
  * Esthesioneuroblastoma
  * CNS lymphoma (primary or systemic disease)
* Multifocal intracranial disease allowed
* No extraneural metastases (except controlled systemic lymphoma)
* Pretreatment considerations based on tumor type

  * Anaplastic astrocytoma:

    * Recurrent disease
    * Any treatment at diagnosis allowed (carmustine dose limited to 480 mg/m2)
    * Chemotherapy not required at recurrence
  * Oligodendroglioma:

    * Disease response (at least minor) to conventional chemotherapy OR
    * Recurrent disease
  * Esthesioneuroblastoma:

    * Attempted complete surgical resection
    * Disease progression after radiotherapy
    * Response to chemotherapy regimen comprising cyclophosphamide, etoposide, and cisplatin
  * CNS lymphoma:

    * Disease refractory to methotrexate OR
    * Failure after initial treatment with methotrexate OR
    * Considered at high risk for disease relapse despite initial response
* Radiographic or pathological confirmation of recurrent disease required
* Not eligible for other high priority national or institutional clinical studies

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG or Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* LVEF at least 45%

Pulmonary:

* DLCO at least 60% predicted OR
* Approval of pulmonologist

Other:

* Not pregnant or nursing
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy
* No concurrent steroids as antiemetics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No concurrent barbiturates or acetaminophen
* Participation in other concurrent supportive care or gene therapy trials allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-04; Primary Completion 2005-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Response rate
Disease-free suvival
Overall survival
Toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States